CLINICAL TRIAL: NCT06897163
Title: A New Method for Ileostomy Output Collection Using an Intestinal Tampon: An Extended Study
Brief Title: A New Method for Ileostomy Output Collection Using an Intestinal Tampon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ampa Medical (Industry)
Responsible Party: Principal Investigator, Cecilie Ammitzbøll, Medical doctor (MD, PhD), Ampa Medical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-23000001
Record Dates: First submitted 2025-01-20; First posted 2025-03-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Ileostomy - Stoma
Keywords: Ileostomy; Stoma care; Stoma management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Specialized Absorbent Intestinal Tampon Group (Experimental): Participants in this arm will receive the specialized absorbent intestinal tampon designed to collect ileostomy output. The study will evaluate the feasibility, safety, and user acceptance of the tampon.
  Interventions: Device: Specialized Absorbent Intestinal Tampon

INTERVENTIONS:
Device: Specialized Absorbent Intestinal Tampon — The specialized absorbent intestinal tampon is designed to be self-inserted by participants with ileostomies. It aims to collect ileostomy output and improve the quality of life by reducing complications associated with traditional stoma bags. The study will test different tampon designs and coatings to find the most suitable one for insertion and retention. Participants will be observed and interviewed during the insertion process, and their feedback on discomfort or pain will be collected using a numerical rating scale (NRS). Stool samples will be collected before and after tampon use for microbiota analysis.

SUMMARY:
The goal of this interventional study is to learn if a specialized absorbent intestinal tampon can effectively collect ileostomy output. The main questions it aims to answer are:

* Can participants successfully self-insert the intestinal tampon?
* What is the level of discomfort or pain associated with the insertion and use of the tampon?

Researchers will compare different tampon designs and coatings to find the most suitable one for insertion and retention. Participants will:

* Be observed and interviewed during the insertion of the tampon by a medical consultant.
* Self-insert the tampon under supervision and later independently.
* Provide feedback on their experience, including any discomfort or pain using a numerical rating scale (NRS).
* Provide stool samples before and after using the tampon for microbiome analysis.

This study aims to determine the feasibility and user acceptance of the intestinal tampon as an alternative to traditional stoma bags, potentially reducing complications and improving the quality of life for people with an ileostomy.

DETAILED DESCRIPTION:
Study Overview This study aims to evaluate the feasibility and user acceptance of a specialized absorbent intestinal tampon designed to collect ileostomy output. The study seeks to address the limitations and complications associated with traditional stoma bags, which have been the standard solution since the 1950s.

Background and Rationale Approximately 1 million people worldwide live with an ileostomy, relying on stoma bags to collect liquid stool. Despite innovations in materials and design, stoma bags still cause significant physical and mental discomfort. Issues include the unsightly appearance of the bag, leakage, noise, and skin irritation. These problems can lead to a reduced quality of life and increased healthcare costs due to skin complications.

The specialized absorbent intestinal tampon is hypothesized to be a discreet and effective alternative to stoma bags. It is designed to be self-inserted by the user, absorb liquid stool, and reduce the complications associated with stoma bags. Previous studies have shown that the tampon can be safely inserted by a healthcare professional, and this study aims to determine if users can safely and effectively insert the tampon themselves.

Study Design and Methods The study is a continuation of a proof-of-concept trial with a qualitative design. It involves observing and interviewing participants during the insertion of the tampon, both by a medical consultant and by the participants themselves. The study will test different tampon designs and coatings to find the most suitable one for insertion and retention.

Participants:

10 individuals with ileostomies, previously screened and included in the study. Inclusion criteria: Age ≥ 18 years, ileostomy > 6 months old, written informed consent, stoma opening ≥ 10 mm in diameter.

Exclusion criteria: Difficulty understanding study information, somatic illness, active inflammatory bowel disease, hernia around the stoma, daily output > 2 liters, active inflammation in the ileum.

Procedures:

Day 1:

Participants arrive at the study site. A medical consultant inserts the tampon and observes the participant. Participants then self-insert the tampon under supervision. The procedure is repeated with different tampon designs, up to three times.

Day 2:

Participants self-insert the tampon using the best method from Day 1. Stool samples are collected before and after tampon use for microbiota analysis.

Participants are interviewed about their experience, including any discomfort or pain using a numerical rating scale (NRS).

The tampon remains in place for up to 6 hours, with participants free to move and eat.

The tampon is removed, and another stool sample is collected. Further testing and iterations may be conducted at home with detailed documentation and follow-up interviews.

Data Collection:

Qualitative data from interviews and observations. Quantitative data from NRS scores for pain and discomfort. Microbiota analysis of stool samples before and after tampon use.

Risks and Benefits The study aims to minimize any discomfort or complications associated with the tampon. Previous safety data indicate no serious risks, but participants are trained and supervised during insertion. Potential risks include pain during insertion, expansion, or removal of the tampon, and rare complications such as tampon retention or perforation.

The potential benefits of the study are significant, as the tampon could provide a more discreet and comfortable alternative to stoma bags, improving the quality of life for individuals with ileostomies.

Ethical Considerations The study adheres to ethical guidelines, including informed consent, data protection, and participant safety. Results will be published in a peer-reviewed journal and on the sponsor's website, regardless of the outcome.

Conclusion This study aims to provide valuable insights into the feasibility and user acceptance of a specialized absorbent intestinal tampon for ileostomy patients. By addressing the limitations of traditional stoma bags, the tampon has the potential to significantly improve the quality of life for individuals with ileostomies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ileostomy > 6 months old
* Stoma opening ≥ 10 mm in diameter
* Written informed consent

Exclusion Criteria:

* Difficulty understanding study information, including language barriers
* Somatic illness, including active inflammatory bowel disease
* Hernia around the stoma
* Daily output > 2 liters
* Active inflammation in the ileum (diagnosed within 2 months before the study day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Self-Insertion of the Intestinal Tampon | Day 1 and Day 2 of the study
  This measure will assess the feasibility of self-inserting the specialized absorbent intestinal tampon. Feasibility will be determined by the percentage of successful insertions, as well as participant feedback and medical consultant observations, which will be reported separately.

SECONDARY OUTCOMES:
Level of Discomfort or Pain During Insertion and Use | Day 2 of the study
  This measure will evaluate the level of discomfort or pain experienced by participants during the insertion and use of the intestinal tampon. Participants will rate their pain using a numerical rating scale (NRS) from 0 to 10.
Changes in Microbiota Composition | Before and after tampon use on Day 2
  This measure will analyze changes in the microbiota composition of stool samples collected before and after using the intestinal tampon. The analysis will focus on the relative abundance of different bacterial species.

CONTACTS AND LOCATIONS:
Locations (1):
- Ampa Medical, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No